CLINICAL TRIAL: NCT04063956
Title: The Efficacy of COGnitive tRaining in patiEnts With Amnestic Mild coGnitive impairmENT (COG-REAGENT): a Multi-center Randomized Controlled Trial
Brief Title: COG-REAGENT: COGnitive tRaining in patiEnts With Amnestic Mild coGnitive impairmENT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xuanwu Hospital, Beijing (Other)
Collaborators: The First Affiliated Hospital of Shanxi Medical University (Other); Shandong Provincial Hospital (Other Government); First Affiliated Hospital of Zhejiang University (Other); The First Hospital of Jilin University (Other); Beijing Friendship Hospital (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); Wuhan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2019042-XZ1
Record Dates: First submitted 2019-08-19; First posted 2019-08-21 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2022-07

CONDITIONS: Amnestic Mild Cognitive Impairment

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive training group (Experimental): Multi-domain adaptive internet-based training program, including processing speed, attention, long-term memory, working memory, flexibility, calculation, and problem solving. 4 x 40 minutes per week, for 12 weeks.
  Interventions: Behavioral: multi-domain internet-based adaptive training program
- Active-control group (Active Comparator): Fixed, primary difficulty level tasks. 4 x 40 minutes per week, for 12 weeks.
  Interventions: Behavioral: active-control program

INTERVENTIONS:
Behavioral: multi-domain internet-based adaptive training program — The training paradigms include a time perception task, visual search task, rapid serial presentation task, delayed match to sample task, paired-associate recall task, attention span task, digit span task, go-no go task, Stroop task, task switching, auditory span task and n-back working memory task. Each task has several difficulty levels. The tasks are grouped in different cognitive domains including: processing speed, attention, perception, long-term memory, working memory, calculation, executive control, reasoning, and problem-solving. Participants in the cognitive training group will complete 40 min of training daily, 4 days a week for 12 weeks. When a high accuracy (80%) is achieved for each task, the level of difficulty will be upgraded for that task.
  Arms: Cognitive training group
Behavioral: active-control program — For the control group, tasks for processing speed and attention are included. Importantly, a fixed, primary difficulty level for all participants in the control group is set.
  Arms: Active-control group

SUMMARY:
This study evaluates the efficacy and mechanism of internet-based cognitive training in patients with amnestic mild cognitive impairment (aMCI). Half of participants will receive multi-domain adaptive internet-based training program, while the other half will receive a fixed, primary difficulty level task.

DETAILED DESCRIPTION:
Background: Alzheimer's disease (AD) is the most common dementia and the major cause for senile dementia. With the increase of life expectancy, AD has become a global problem. However, to date, drug therapies only have modest benefits for patients with AD. Recently, researchers have begun to focus on early intervention of AD at its preclinical stages. Individuals with amnestic mild cognitive impairment (aMCI), often the prodromal stage of AD, report mild short-term memory difficulties but preserved independence in activities of daily living. The aMCI stage is important to slow or even prevent the development of AD. Some previous studies have suggested cognitive training is a potential non-pharmacological intervention for aMCI, however, the results were inconsistent. Thus, investigators will conduct this multi-center randomized controlled trial to explore whether and how cognitive training improves cognitive function in patients with aMCI.

Objectives: The first aim of this multi-center single-blinded, randomized controlled trial is to assess whether internet-based cognitive training improves cognitive abilities in patients with aMCI. Furthermore, the second objective is to evaluate the effect of cognitive training on neural plasticity, including brain activation and white matter integrity, which are assessed by functional and structural MRI.

Patients and Methods: The study will include 260 patients diagnosed with aMCI from eight centers around China. The patients will be randomized to either a cognitive training group or an active-control group. The intervention is 12-week internet-based cognitive training performed for 40 minutes per day, 4 days a week. Within each task, high accuracy (80%) is required to upgrade to the next difficulty level. The active- control group will receive five processing speed and attention tasks, whose duration also total to 40 min each training day. However, these tasks are set to a fixed, primary difficulty level across the study.

Neuropsychological assessments and structural and functional magnetic resonance imaging (MRI) will be performed at the baseline, end of intervention, and 6 months after randomization to measure long-term resilience of the effect.

Relevance: Early intervention of aMCI has the potential to delay or even prevent the development of dementia. Some previous studies have suggested cognitive training is a potential non-pharmacological intervention for aMCI, however, the results were inconsistent. Thus, the proposed study is to determine the efficacy of cognitive training in patients with aMCI. Secondly, using functional and structural MRI, this study is to reveal the potential mechanisms underlying cognitive training.

ELIGIBILITY:
Inclusion Criteria:

1. Literate Han Chinese, 50-85 years of age with a caregiver that accompanies the subject consistently at least 4 days a week;
2. Complaint and/or informant report of a cognitive impairment lasting for at least 3 months;
3. Clinical diagnosis of MCI according to the MCI core clinical criteria of the National Institute on Aging-Alzheimer's Association (NIA-AA) guidelines;
4. A prominent manifestation of memory deficit with or without other cognitive domain impairments;
5. Mini-Mental State Examination (MMSE) score ≥24, and Clinical dementia rating (CDR) = 0.5, and
6. Normal or slightly impaired activities of daily living as defined by a total score of ≤ 1.5 on the three functional CDR domains (home and hobbies, community affairs, and personal care).

Exclusion Criteria:

1. Severe aphasia, physical disabilities, or any other disease that may preclude completion of neuropsychological testing;
2. A medical history of stroke with focal neurological features including hemiparesis, sensory loss, visual field deficits, and evidence of responsible lesions on MRI;
3. Significant white matter lesions (Fazekas score = 3-6);
4. Disorders other than aMCI that may affect cognition;
5. Depression or other psychiatric disorders;
6. Clinically significant gastrointestinal, renal, hepatic, respiratory, infectious, endocrine, or cardiovascular diseases, cancer, alcoholism, drug addiction;
7. Use of medications that may affect cognitive functioning, including tranquilizers, anti-anxiolytics, hypnotics, nootropics, and cholinomimetic agents;
8. Inability to undergo a brain MRI; and
9. Other conditions that in the investigator's opinion might not be suitable for the study.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2019-11-06 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Change in Montreal Cognitive Assessment | 12 weeks (end of intervention)
  Montreal Cognitive Assessment (MoCA) will be used to evaluate the general cognitive function. MoCA ranges from 0 to 30, and higher value represents a better outcome.

SECONDARY OUTCOMES:
Change in Alzheimer's Disease Assessment Scale cognitive subscale (ADAS-cog, 11-items version). | 12 weeks (end of intervention), 6 months
  ADAS-cog 11 scale ranges from 0 to 70, and higher value represents a worse outcome. This study will use ADAS-cog to assess changes in the global cognitive function after intervention.
Change in brain volume and white matter integrity | 12 weeks (end of intervention), 6 months
  Structural MRI will be used to measure brain volume and white matter integrity.
Change in brain connectivity | 12 weeks (end of intervention), 6 months
  Functional MRI will be used to measure brain connectivity.
Change in Mini-mental State Examination | 12 weeks (end of intervention), 6 months
  Mini-mental State Examination (MMSE) will be used to evaluate the general cognitive function. MMSE ranges from 0 to 30, and higher value represents a better outcome.
Change in Montreal Cognitive Assessment | 6 months
  Montreal Cognitive Assessment (MoCA) will be used to evaluate the general cognitive function. MoCA ranges from 0 to 30, and higher value represents a better outcome.
Change in memory function | 12 weeks (end of intervention), 6 months
  WHO-UCLA Auditory Verbal Learning Test will be used to assess memory function. It ranges from 0 to 45, and higher value represents a better outcome.
Change in Digit span forward | 12 weeks (end of intervention), 6 months
  Digit span will be used to assess attention. It ranges from 3 to 10, and higher value represents a better outcome.
Change in Digit span backward | 12 weeks (end of intervention), 6 months
  Digit span backward will be used to assess executive function. It ranges from 2 to 8, and higher value represents a better outcome.
Change in Trail Making Test | 12 weeks (end of intervention), 6 months
  Trail-Making Test B minus A score will be used to assess executive function. Trail-Making Test B minus A ranges from -150 to 300, higher value represents a worse outcome.
Change in Boston Naming Test | 12 weeks (end of intervention), 6 months
  Boston Naming Test will be used to assess language function. It ranges from 0 to 30, and higher value represents a better outcome.
Change in Activities of Daily Living | 12 weeks (end of intervention), 6 months
  Activities of Daily Living (ADL) scale will be used to assess the change of life quality. It ranges from 20 to 80. The "20" represents normal life ability and the higher score presents the worse life ability.
Change in Clinical Dementia Rating Scale sum of the boxes | 12 weeks (end of intervention), 6 months
  Clinical Dementia Rating Scale sum of the boxes (CDR-SB) will be used to evaluate the general cognitive function. CDR-SB ranges from 0 to 18, and higher value represents a worse outcome.
Change in Quality of Life-Alzheimer's Disease (QoL-AD) Scale | 12 weeks (end of intervention), 6 months
  Quality of Life-Alzheimer's Disease (QoL-AD) Scale will be used to evaluate the life quality of the patients. The total score is 13-52, with higher scores indicating better QoL.
Change in Cookie Theft picture description task | 12 weeks (end of intervention), 6 months
  Cookie Theft picture description task will be used to evaluate spontaneous discourse. We will analyze the total number of syllables produced, the total number of information units produced, and the total time taken to describe the picture

CONTACTS AND LOCATIONS:
Overall Officials: Yi Tang, M.D., Ph.D., Principal Investigator — Xuanwu Hospital, Beijing
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, China

REFERENCES:
- [Derived] Xing Y, Zhu Z, Du Y, Zhang J, Qu Q, Sun L, Li Y, Guo Y, Peng G, Liu Y, Yu Y, Qiao Y, Xie B, Shi X, Lu J, Jia J, Tang Y. The Efficacy of COGnitive tRaining in patiEnts with Amnestic mild coGnitive impairmENT (COG-REAGENT): Protocol for a Multi-Center Randomized Controlled Trial. J Alzheimers Dis. 2020;75(3):779-787. doi: 10.3233/JAD-191314. PMID 32333590